CLINICAL TRIAL: NCT05874297
Title: Feasibility and Pilot Study Testing an Online Digital Intervention to Improve Symptom Management During Breast Cancer Chemotherapy
Brief Title: Online Nutrition Education to Decrease the Side Effects of Chemotherapy in Patients With Breast Cancer
Acronym: ONE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1122898; NCI-2022-10270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11109 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-12-20; First posted 2023-05-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): Patients receive standard of care consisting of symptom monitoring, scheduled nurse visits, and access to current Cook for Your Life website.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (enhanced Cook for Your Life) (Experimental): Patients receive standard of care as in Arm I and access to enhanced Cook for Your Life information on symptom management.
  Interventions: Behavioral: Internet-Based Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm I (standard of care)
Behavioral: Internet-Based Intervention — Access to enhanced Cook for your life website
  Arms: Arm II (enhanced Cook for Your Life)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial tests an online nutrition education program focused on decreasing nutrition-related side effects of chemotherapy in patients with breast cancer. Patients undergoing chemotherapy are at risk for complications such as diarrhea or constipation which can lead to poor nutritional intake and malabsorption of nutrients. This study is testing the effects of information delivered via the Cook for Your Life website in conjunction with standard clinical care to improve symptom management during chemotherapy treatment for breast cancer, which could serve as a new model for supportive oncology care.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care consisting of symptom monitoring, scheduled nurse visits, and access to current Cook for Your Life website.

ARM II: Patients receive standard of care as in Arm I and access to enhanced Cook for Your Life information on symptom management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Stage I-III breast cancer.
* Current breast cancer patients scheduled to receive ddAC-T(+/-C), TCHP, or TCPembro-AC chemotherapy at Fred Hutch South Lake Union (can enroll prior to receipt of 2nd cycle).
* Not pregnant and no plan to become pregnant during chemotherapy treatment.
* Ability to speak and read English.
* Access to smartphone, tablet, or computer and Internet.
* Willing and able to complete all study activities through the end of chemotherapy, including completing online questionnaires and telephone assessments.
* Women must not be pregnant at time of enrollment based on self-report.
* Able to understand and willing to sign written informed electronic (e) consent in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Accrual rate | ~4 months
  Accrual rate to the study.
Use of cook for your life website pages (adherence: visiting website) will be measured via Google analytics | ~4 months
  Google analytics will be used to identify whether participants visit the website.
Use of cook for your life website pages (adherence: webpages viewed) will be measured via Google analytics | ~4 months
  Google analytics will be used to identify what webpages participants view.
Time of use of cook for your life website (adherence: total time) will be measured via Google analytics | ~4 months
  Google analytics will be used to measure how much total time spent on the website.
Time of use of cook for your life website (adherence: time per webpage) will be measured via Google analytics | ~4 months
  Google analytics will be used to measure time spent per webpage visited.
User pathways of cook for your life website (adherence) will be measured via Google analytics | ~4 months
  Google analytics will be used to determine the order/sequence of webpages participants follow to navigate through the website.
Participant retention will be measured via participants competing surveys at all timepoints | ~4 months
  The number of participants who complete all study activities through the end of chemotherapy.
Acceptability of cook for your life website will be measured via an exit interview | ~4 months
  Participant acceptability of cook for your life website will be assessed via a short semi-structured exit interview.

SECONDARY OUTCOMES:
Incidence of patient-reported nutrition-related adverse events | ~4 months
  Patient-reported nutrition-related adverse events assessed via the chemotherapy patient reported outcome (PRO) tool.
Number of participants with treatment delays and causes of delays | ~4 months
  Treatment delays and causes of delays as assessed via chart abstraction
Delivered dose of planned treatment | ~4 months
  Assessed via chart abstraction.
Change in dose | ~4 months
  Assessed via chart abstraction.
Change in weight | ~4 months
  Weight change as assessed via chart abstraction.
Medication adherence assessed via chart abstraction | ~4 months
  Participant medication usage assessed via chart abstraction to note medications including anti-emetics, proton pump inhibitors, anti-depressants, and anti-anxiety medication.
Quality of life as assessed via The Patient-Reported Outcome Measurement Information System (PROMIS)-Global | ~4 months
  The PROMIS Global scale contains 10 items that measure self-reported physical, mental, and social health. Each question is scored on a 1 - 5 scale with a total score range of 4 - 20. Higher scores indicate better overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No